CLINICAL TRIAL: NCT01119222
Title: A Randomised, Double-Blind, Double-Dummy, Placebo And Active Controlled, 4-Way Crossover Methodology Study To Assess The Effect Of Gabapentin, Diphenhydramine And Morphine On Cold Pain In Healthy Male Volunteers
Brief Title: Study To Assess The Effect Of Gabapentin, Diphenhydramine And Morphine On Cold Pain In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: A9001388
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Results first posted 2011-03-07 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: Cold pain methodology; Healthy male volunteers; gabapentin; Diphenhydramine; morphine
MeSH Terms: interventions — Gabapentin; Diphenhydramine; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Gabapentin 1200mg (Active Comparator)
  Interventions: Drug: Gabapentin
- Diphenhydramine 50 mg (Active Comparator)
  Interventions: Drug: Diphenhydramine
- Morphine 10 mg (Active Comparator)
  Interventions: Drug: Morphine
- Placebo formulations (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Capsule, single 1200mg dose
  Arms: Gabapentin 1200mg
Drug: Diphenhydramine — Tablet, single 50mg dose
  Arms: Diphenhydramine 50 mg
Drug: Morphine — IV, single 10mg dose
  Arms: Morphine 10 mg
Drug: Placebo — Placebo formulations (Capsule, tablet, IV to match the active treatments and to be administered in a double-dummy fashion).
  Arms: Placebo formulations

SUMMARY:
Human experimental pain models are useful in understanding the mechanisms underlying clinical pain conditions and can be used to test the analgesic efficacy of drugs used in the management of pain. Once established these models can be used as mechanism biomarkers in early development clinical studies to establish proof of mechanism for novel compounds. The cold pain model is a mechanistic pain biomarker with potential application in proof of mechanism studies. In this study we aim to set up this cold pain model at a Clinical Research Unit and demonstrate we can effectively screen subjects for this model and examine the effect of morphine, diphenhydramine, and gabapentin in the cold pain model.

DETAILED DESCRIPTION:
Cold pain methodology development

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers having given consent to participate in the study who have no clinically significant anomalies and whose vital signs are within normal range.
* Subject having performed the cold pain test reproducibly ie, if the area under the pain-time curve (AUC) must be within 20% during successive tests within one cold pain test screening visit and within 30% between the two cold pain test screening visits.

Exclusion Criteria:

* Subject who have had a serious adverse reaction or significant hypersensitivity to any of the study drugs.
* Subjects with a history of or evidence of any neurological condition which could affect pain sensation.
* Subjects with an AUCcpt 0-120 sec in the cold pain test of <1000 in any of the screening tests (excluding familiarization).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001388&StudyName=Study%20To%20Assess%20The%20Effect%20Of%20Gabapentin%2C%20Diphenhydramine%20And%20Morphine%20On%20Cold%20Pain%20In%20Healthy%20Male%20Volunteers

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to entering the treatment phases of the study, participants were required to successfully pass cold pain screening tests. Twenty participants were randomized and 19 participants received treatment consisting of a crossover sequence of 4 study drugs administered in sequence I, II, III or IV.
Groups:
- Placebo, Morphine, Diphenhydramine, Gabapentin: Placebo (capsules, tablet and intravenous (IV) first, then morphine 10 mg IV, then diphenhydramine 50 mg tablet, then gabapentin 1200 mg capsule.
- Morphine, Gabapentin, Placebo, Diphenhydramine: Morphine 10 mg intravenous (IV) first, then gabapentin 1200 mg capsule, placebo (capsules, tablet and IV), then diphenhydramine 50 mg tablet.
- Gabapentin, Diphenhydramine, Morphine, Placebo: Gabapentin 1200 mg capsule first, then diphenhydramine 50 mg tablet, then morphine 10 mg intravenous (IV), then placebo (capsules, tablet and IV).
- Diphenhydramine, Placebo, Gabapentin, Morphine: Diphenhydramine 50 mg tablet first, then placebo (capsules, tablet and intravenous (IV), then gabapentin 1200 mg capsule, then morphine 10 mg IV.
Period: Overall Study
Arm/Group | Placebo, Morphine, Diphenhydramine, Gabapentin | Morphine, Gabapentin, Placebo, Diphenhydramine | Gabapentin, Diphenhydramine, Morphine, Placebo | Diphenhydramine, Placebo, Gabapentin, Morphine
Started | 5 | 5 | 5 | 4
Completed | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all participants who initiated in any treatment sequence
Arm/Group | Entire Study Population
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Average Pain (0-120 Seconds): Cold Pain Test Visual Analog Scale (VAS)
Description: Area under the cold pain test Visual Analog Scale (VAS) time curve (AUCcpt 0 to 120 seconds [sec]) averaged over the 120 sec for each time point assessed. Participant adjusted 100 millimeter (mm) electronic VAS with range of "no pain" (0) to "maximum pain" (100) at the anchor endpoints of the scale and "moderate pain" at the midpoint. Pain reported while non-dominant hand was placed in thermostatically controlled water bath at 2±1°C for a maximum of 120 sec.
Time Frame: Pre-dose, 1, 1.5, 2, 4, and 8 hours post-dose
Population: Participants for analysis = participants who completed all of the four treatment periods.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Gabapentin: Gabapentin single oral 1200 mg dose
- Morphine: Morphine single IV 10 mg dose
- Diphenhydramine: Diphenhydramine single oral 50 mg dose
- Placebo: Oral and IV doses to match active treatments
Arm/Group | Gabapentin | Morphine | Diphenhydramine | Placebo
Number analyzed (Participants) | 19 | 19 | 19 | 19
mm
  Pre-dose | 45.2 (16.15) | 45.5 (16.10) | 45.0 (16.66) | 44.9 (15.16)
  1 hour | 41.9 (16.95) | 28.6 (16.88) | 45.1 (17.29) | 38.4 (15.69)
  1.5 hours | 39.4 (16.21) | 26.1 (18.28) | 42.3 (16.67) | 40.2 (17.75)
  2 hours | 40.4 (17.71) | 25.6 (18.44) | 40.5 (17.22) | 39.5 (16.86)
  4 hours | 41.9 (16.37) | 34.7 (18.29) | 44.2 (17.35) | 44.3 (16.70)
  8 hours | 44.7 (15.06) | 36.7 (17.14) | 43.8 (15.08) | 44.2 (14.55)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Pre-dose; mixed effect model with random subject effect, fixed period and treatment effects and random subject-by-visit effect as residual. Sample sizing calculated based on results from previous methodology studies performed using the same cold pain test; primary criteria was ability to detect a significant gabapentin effect over placebo; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.28, 90% CI 2-sided [-3.82 to 4.38], Standard Error of Mean 2.45
Statistical Analysis 2: Comparison: Morphine vs Placebo; Pre-dose; mixed effect model with random subject effect, fixed period and treatment effects and random subject-by-visit effect as residual; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.58, 90% CI 2-sided [-3.53 to 4.68], Standard Error of Mean 2.45
Statistical Analysis 3: Comparison: Diphenhydramine vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 90% CI 2-sided [-3.99 to 4.22], Standard Error of Mean 2.45
Statistical Analysis 4: Comparison: Gabapentin vs Placebo; 1 hour post-dose: mixed effect model with random subject effect, fixed period and treatment effects and random subject-by-visit effect as residual; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.14, 90% CI 2-sided [-1.15 to 5.44], Standard Error of Mean 1.97
Statistical Analysis 5: Comparison: Morphine vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -11.18, 90% CI 2-sided [-14.48 to -7.89], Standard Error of Mean 1.97
Statistical Analysis 6: Comparison: Diphenhydramine vs Placebo; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 5.49, 90% CI 2-sided [2.20 to 8.78], Standard Error of Mean 1.96
Statistical Analysis 7: Comparison: Gabapentin vs Placebo; 1.5 hours post-dose: mixed effect model with random subject effect, fixed period and treatment effects and random subject-by-visit effect as residual; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.73, 90% CI 2-sided [-5.53 to 4.08], Standard Error of Mean 2.87
Statistical Analysis 8: Comparison: Morphine vs Placebo; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -13.93, 90% CI 2-sided [-18.74 to -9.13], Standard Error of Mean 2.87
Statistical Analysis 9: Comparison: Diphenhydramine vs Placebo; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.88, 90% CI 2-sided [-2.01 to 7.78], Standard Error of Mean 2.92
Statistical Analysis 10: Comparison: Gabapentin vs Placebo; 2 hours post-dose: mixed effect model with random subject effect, fixed period and treatment effects and random subject-by-visit effect as residual; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.82, 90% CI 2-sided [-5.32 to 6.96], Standard Error of Mean 3.66
Statistical Analysis 11: Comparison: Morphine vs Placebo; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -13.12, 90% CI 2-sided [-19.14 to -7.09], Standard Error of Mean 3.59
Statistical Analysis 12: Comparison: Diphenhydramine vs Placebo; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.58, 90% CI 2-sided [-4.45 to 7.60], Standard Error of Mean 3.59
Statistical Analysis 13: Comparison: Gabapentin vs Placebo; 4 hours post-dose: mixed effect model with random subject effect, fixed period and treatment effects and random subject-by-visit effect as residual; Test type: Superiority or Other; Mean Difference (Final Values) = -2.53, 90% CI 2-sided [-7.39 to 2.32], Standard Error of Mean 2.90
Statistical Analysis 14: Comparison: Morphine vs Placebo; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -9.59, 90% CI 2-sided [-14.44 to -4.73], Standard Error of Mean 2.90
Statistical Analysis 15: Comparison: Diphenhydramine vs Placebo; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.00, 90% CI 2-sided [-4.85 to 4.85], Standard Error of Mean 2.90
Statistical Analysis 16: Comparison: Gabapentin vs Placebo; 8 hours post-dose: mixed effect model with random subject effect, fixed period and treatment effects and random subject-by-visit effect as residual; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.49, 90% CI 2-sided [-3.23 to 4.22], Standard Error of Mean 2.22
Statistical Analysis 17: Comparison: Morphine vs Placebo; [analysis description as in outcome 1, analysis 16]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -7.47, 90% CI 2-sided [-11.19 to -3.75], Standard Error of Mean 2.22
Statistical Analysis 18: Comparison: Diphenhydramine vs Placebo; [analysis description as in outcome 1, analysis 16]; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.27, 90% CI 2-sided [-3.99 to 3.45], Standard Error of Mean 2.22

2. Primary Outcome: Interpolated Average Pain (0-8 Hours)
Description: Interpolated average pain (0 to 8 hours): area under the curve (AUC) of average pain (0 to 120 seconds) recorded at each of the time points taken over 8 hour time period divided by 8.
Time Frame: Pre-dose to 8 hours post-dose
Population: Participants for analysis = participants who completed all of the four treatment periods.
Measure: Least Squares Mean (Standard Error); unit: hours
Groups:
- Gabpentin: Gabapentin 1200 mg
- Morphine: Morphine 10 mg
Arm/Group | Gabpentin | Morphine | Diphenhydramine | Placebo
Number analyzed (Participants) | 19 | 19 | 19 | 19
hours | 42.2 (3.67) | 33.4 (3.67) | 43.6 (3.67) | 42.8 (3.67)
Statistical Analysis 1: Comparison: Gabpentin vs Placebo; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.60, 90% CI 2-sided [-4.24 to 3.04], Standard Error of Mean 2.17
Statistical Analysis 2: Comparison: Morphine vs Placebo; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -9.43, 90% CI 2-sided [-13.07 to -5.79], Standard Error of Mean 2.17
Statistical Analysis 3: Comparison: Diphenhydramine vs Placebo; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.84, 90% CI 2-sided [-2.80 to 4.48], Standard Error of Mean 2.17

3. Secondary Outcome: Number of Participants With Clinically Significant Findings in Vital Signs
Description: Supine blood pressure measured to nearest millimeter of mercury (mmHg), pulse rate measured with automated device or manually in the brachial/radial artery for at least 30 seconds.
Time Frame: Predose, Day 1, Day 2 each treatment period, follow-up visit (at least 7 days after last dosing)
Population: Safety population: all subjects who received at least 1 dose of study medication. Although individual listing data for vital signs were collected, summary statistics were not generated for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Gabapentin | Morphine | Diphenhydramine | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Findings on Physical Examination
Description: Full physical examination consisting of an examination of the abdomen, cardiovascular systems, lungs, lymph nodes, mouth, musculoskeletal and neurological systems, skin, extremities, head, ears, eyes, nose, throat and thyroid gland.
Time Frame: Pre-dose and follow-up visit (at least 7 days after last dosing)
Population: Safety population: all subjects who received at least 1 dose of study medication. Although individual subject data were collected, results were not captured for inclusion in the study database.
Measure: Number; unit: participants
Arm/Group | Gabapentin | Morphine | Diphenhydramine | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Abnormal Findings on Electrocardiogram (ECG)
Description: Standard 12-lead ECG performed after subject had rested quietly for at least 10 minutes in a supine position.
Time Frame: Pre-dose and follow-up visit (at least 7 days after last dosing)
Population: Safety population: all subjects who received at least 1 dose of study medication. Although individual subject data were collected and monitored, summary statistics were not generated for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Gabapentin | Morphine | Diphenhydramine | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormal Haematology, Clinical Chemistry, Urinalysis Results
Description: Standard haematology, clinical chemistry, and urinalysis safety laboratory tests.
Time Frame: Pre-dose, follow-up visit (at least 7 days after last dosing)
Population: as for outcome 5
Measure: Number; unit: particpants
Groups:
- Gabapentin: Gabapentin 1200 mg
Arm/Group | Gabapentin | Morphine | Diphenhydramine | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormal Cardiac Monitoring Results
Description: Continuous cardiac monitoring during intervenous (IV) infusion dosing (morphine or placebo).
Time Frame: Pre-dose through duration of IV infusion dosing
Population: Safety population: all subjects who received at least 1 dose of study medication. Although continuous cardiac monitoring was performed throughout IV dosing, results were not captured for inclusion in the study database.
Measure: Number; unit: participants
Arm/Group | Gabapentin | Morphine | Diphenhydramine | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Abnormal Pulse Oxymetry Results
Description: Pulse oxymetry to monitor percentage of hemoglobin saturated with oxygen during intervenous (IV) infusion dosing (morphine or placebo).
Time Frame: Predose through duration of IV infusion dosing
Population: Safety population: all subjects who received at least 1 dose of study medication. Although pulse oxymetry was performed throughout IV dosing, results were not captured for inclusion in the study database.
Measure: Number; unit: participants
Arm/Group | Gabapentin | Morphine | Diphenhydramine | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Safety population: all subjects who received at least 1 dose of study medication. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Gabapentin | Morphine | Diphenhydramine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 9/19 | 18/19 | 5/19 | 3/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin (N=19) | Morphine (N=19) | Diphenhydramine (N=19) | Placebo (N=19)
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 7 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 3 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 2
Feeling abnormal (General disorders) | 2 | 7 | 0 | 0
Feeling drunk (General disorders) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 1 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 4 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 4 | 0 | 0
Somnolence (Nervous system disorders) | 6 | 7 | 5 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Stress (Psychiatric disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.